CLINICAL TRIAL: NCT05423379
Title: XIENCE Skypoint Large Vessel Post Approval Study
Acronym: SPIRIT XLV PAS
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT -CIP 10445
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: ABT -CIP 10445; Coronary artery disease; XIENCE; Large Vessel; Skypoint
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- XIENCE Skypoint Large Vessel Everolimus Eluting Coronary Stent System: Subjects who were implanted with XIENCE Skypoint Large Vessel Everolimus Eluting Coronary Stent System will be included.
  Interventions: Device: XIENCE Skypoint Large Vessel Everolimus Eluting Coronary Stent System (EECSS)

INTERVENTIONS:
Device: XIENCE Skypoint Large Vessel Everolimus Eluting Coronary Stent System (EECSS) — XIENCE Skypoint Large Vessel EECSS is composed of a L-605 CoCr stent and coated with poly (n-butyl methacrylate) (PBMA) primer and a drug coating formulation of polymer of vinylidene fluoride and hexafluoropropylene (PVDF-HFP)/everolimus pre-mounted on a balloon catheter delivery system.

SUMMARY:
SPIRIT XLV PAS is a prospective, single arm, multi-center, US and OUS post-approval observational study to evaluate the continued safety and effectiveness of the XIENCE Skypoint Large Vessel Everolimus Eluting Coronary Stent System (EECSS) Large Vessel (LV) sizes (diameter 4.5 mm and 5.0 mm) during commercial use in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent per site requirements.
3. Subject must have evidence of myocardial ischemia (STEMI, NSTEMI, Unstable Angina or Stable Angina) or who have silent ischemia with evidence of ischemia, appropriate for PCI treatment with DES. Subject with stable angina or silent ischemia must have objective sign of ischemia as suggested by one of the following:

   1. Abnormal stress or imaging stress test
   2. Abnormal computed tomography-fractional flow reserve (CT-FFR)
   3. Stenosis by visual estimation ≥ 70%
   4. Abnormal pressure-derived indexes (FFR, instantaneous wave-free ratio [iFR], or relative flow reserve [RFR])
4. Subject must agree not to participate in any other clinical study for a period of one year following the index procedure.

Angiographic Inclusion Criteria

1. Patients who have lesion(s) in a vessel with reference vessel diameter > 4.25 mm and ≤ 5.25 mm as the target lesion
2. Patients who receive at least one Skypoint LV stent

   1. Lesions with RVD ≤ 4.25 mm should be treated as the non-target lesions during the index procedure with commercially available XIENCE family of stents
   2. Up to three lesions (target and non-target) in two coronary vessels can be treated at the index procedure.

Exclusion Criteria:

General Exclusion Criteria

1. Patients who have contraindications of the Skypoint LV per the IFU
2. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the prior 2 months.

Angiographic Exclusion Criteria:

1. Patients who require three vessel treatment.
2. If left main coronary artery (LMCA) is the intended target vessel, patients who have unprotected left main disease with the SYNTAX Score ≥ 23

   1. Unprotected LM disease with a SYNTAX score ≤ 22 (site-assessment) can be treated as the target lesion but not to exceed 40% of the study population
   2. A heart team consensus approach per site's standard of care (SOC) to enhance patient protection and optimal clinical practice for the left main treatment is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of all genders from the general population who have at least one XIENCE Skypoint LV implanted.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Target Lesion Failure (TLF) at 1 year | At 1 Year
  TLF is defined as the composite of cardiac death, myocardial infarction related to the target vessel (TV-MI), or ischemic driven target lesion revascularization (ID-TLR).

CONTACTS AND LOCATIONS:
Locations (18):
- United States (13):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Bryan Heart, Lincoln, Nebraska
  - Lenox Hill Hospital, New York, New York
  - Pinnacle Health System, Wormleysburg, Pennsylvania
  - Anmed Health, Anderson, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Hendrick Medical Center, Abilene, Texas
  - Austin Heart, Austin, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Shannon Clinic, San Angelo, Texas
- France (2):
  - Clinique Pasteur Toulouse, Toulouse, Midi-Pyrenees
  - Hopital Cardiovasculaire et Pneumologique Louis Pradel, Lyon, Rhone
- Spain (3):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen de Rocio, Seville

IPD SHARING:
Plan to Share IPD: Undecided